**Study Title:** Pharmacodynamic Biomarkers to Support Biosimilar Development: Clinical Study 2 (PCSK9 Inhibitors – Alirocumab and Evolocumab)

**Document Title:** Statistical Analysis Plan – Study No. SCR-007

**Document Date: 23 July 2021** 

NCT Number: NCT04189484

## Statistical Analysis Plan

#### SCR-007: Pharmacodynamic Biomarkers to Support Biosimilar Development: Clinical Study 2 (PCSK9 Inhibitors – Alirocumab and Evolocumab)

**Sponsor:** U.S. Food and Drug Administration

White Oak Building #64, Room 2072

10903 New Hampshire Avenue

Silver Spring, MD 20993

**Sponsor Study Lead:** David Strauss, MD, PhD

Director, Division of Applied Regulatory Science

U.S. Food and Drug Administration

Telephone: 301-796-6323

Email: david.strauss@fda.hhs.gov

Sponsor Medical Keith Burkhart, MD

**Monitor:** U.S. Food and Drug Administration

Telephone: 301-796-2226

Email: keith.burkhart@fda.hhs.gov

**Project Manager:** Jeffry Florian, PhD

U.S. Food and Drug Administration

Telephone: 301-796-4847

Email: Jeffry.florian@fda.hhs.gov

**Study Monitor:** Jill Brown

FDA IRB Project Manager

U.S. Food and Drug Administration

Version of SAP: 3.0

**Date of SAP:** July 23, 2021

#### **CONFIDENTIAL**

The concepts and information contained in this document or generated during the study are considered proprietary and may not be disclosed in whole or in part without the expressed written consent of the U.S. Food and Drug Administration.

#### **Sponsor Signatures Page**

#### Prepared by

# Jeffry Florian - S ou=FDA, ou=People, cn=Jeffry Florian - S, ou=FDA, o

Digitally signed by Jeffry Florian -S DN: c=US, o=U.S. Government, ou=HHS, 0.9.2342.19200300.100.1.1=2000498765 Date: 2021.07.25 20:48:08 -04'00'

Jeffry Florian, PhD **Associate Director** Division of Applied Regulatory Science U.S. Food and Drug Administration

Date

#### Reviewed by

Morasa Sheikhy -S (Affiliate)

Digitally signed by Morasa Sheikhy -S (Affiliate) DN: c=US, o=U.S. Government, ou=HHS, ou=FDA, ou=People, 0.9.2342.19200300.100.1.1=2003067248, cn=Morasa Sheikhy -S (Affiliate) Date: 2021.07.26 08:53:09 -04'00'

Morasa Sheikhy, PharmD **ORISE Fellow** Division of Applied Regulatory Science U.S. Food and Drug Administration

Date

Approved by

Digitally signed by David Strauss -S DN: c=US, o=U.S. Government, ou=HHS, ou=FDA, ou=People, cn=David Strauss -S, 0.9.2342.19200300.100.1.1=2000507494 Date: 2021.07.24 19:31:43 -04'00'

David Strauss, MD, PhD

Director

Division of Applied Regulatory Science U.S. Food and Drug Administration

Date

## **Contents**

| Spo | onsor | Signa | itures Page | 2 |
|---|---|---|---|---|
| Tal | ole of | Abbr | eviations | 5 |
| Cha | ange L | ₋og | | 6 |
| 1. | Intr | oduc | tion | 7 |
| 2. | Stud | dy Ol | ojectives | 7 |
| : | 2.1. | Prin | nary Objective | 7 |
| : | 2.2. | Sec | ondary Objectives | 7 |
| : | 2.3. | Exp | loratory Objective | 7 |
| 3. | Stud | dy Ov | verview | 7 |
| 3 | 3.1. | Stud | dy Design | 7 |
| 3 | 3.2. | Sam | nple size | 8 |
| 4. | Stud | dy En | dpoints | 8 |
| 4 | 4.1. | Prin | nary Endpoints | 8 |
| 4 | 4.2. | Sec | ondary Endpoints | 9 |
| 4 | 4.3. | Ехр | loratory Endpoints | 9 |
| 5. | Ana | lysis | Populations | 9 |
| 6. | Data | a Scr | eening and Acceptance | 10 |
| ( | 5.1. | Han | dling of Missing and Incomplete Data | 10 |
| 7. | Gen | eral | Statistical Considerations | 10 |
| - | 7.1. | Sub | ject Disposition | 11 |
| - | 7.2. | Den | nographics and Baseline Characteristics | 11 |
| - | 7.3. | Pha | rmacodynamic Analysis | 11 |
| | 7.3. | 1 | LDL-C | 11 |
| | 7.3. | 2 | ApoB and PCSK9 | 11 |
| - | 7.4. | Pha | rmacokinetic Analysis – Alirocumab and Evolocumab | 12 |
| - | 7.5. | PK/ | PD Analyses | 12 |
| - | 7.6. | Exp | loratory Omics Analysis | 13 |
| - | 7.7. | Safe | ety Analyses | 13 |
| | 7.7. | 1 | Adverse Events | 13 |
| | 7.7. | 2 | Clinical Laboratory Tests | 14 |
| | 7.7. | 3 | Vital Sign Measurements | 14 |

| | 7.7.4 | Safety 12lead Electrocardiograms | 14 |
|---|---|---|---|
| | 7.7.5 | Physical Examinations | 14 |
| | 7.7.6 | Other Safety Data | 14 |
| 8. | Data Qu | ality Assurance | 14 |
| A | tachment A | A. Pharmacokinetic, Pharmacodynamic, and Biomarker Sample Collection Schedule | 16 |
| | Pharmaco | kinetic Sample Collection | 16 |
| | Pharmaco | dynamic Sample Collection | 16 |
| | Explorator | y PD Biomarkers | 16 |
| A | tachment I | 3. Randomization Schedule | 17 |

### **Table of Abbreviation**

| Abbreviation | Definition |
|---|---|
| ApoB | apolipoprotein B |
| $\Delta { m ApoB}_{ m min}$ | maximum decrease from baseline in ApoB |
| $\mathrm{AUC}_{0	ext{-}\mathrm{inf}}$ | area under the concentration-time curve from time zero to infinity |
| $\mathrm{AUC}_{0	ext{-t}}$ | area under the concentration-time curve from time zero to last on-<br>study sample |
| $\mathrm{AUEC}_{0	ext{-t}}$ | area under the effect curve from time zero to last on-study sample |
| AUEC | area under the effect curve |
| $pAUEC_{0-t}$ | percentage area under the effect curve from time zero to last on-<br>study sample |
| CL/F | apparent clearance |
| $C_{max}$ | maximum observed concentration |
| $EC_{50}$ | the exposure that gives-half maximal response, model parameter |
| $ED_{50}$ | the dose that gives-half maximal response, model parameter |
| $E_{\text{max,exp}}$ | maximum PD response, model parameter - concentration analysis |
| $E_{\rm max,dose}$ | maximum PD response, model parameter – dose analysis |
| FDA | Food and Drug Administration |
| $K_{el}$ | elimination rate |
| LDL-C | low-density lipoprotein (LDL) cholesterol |
| $\Delta LDL$ - $C_{min}$ | maximum decrease from baseline in LDL-C |
| mg | Milligram |
| PCSK9 | proprotein convertase subtilisin/kexin type 9 |
| $\Delta PCSK9_{min}$ | maximum decrease from baseline in PCSK9 |
| PD | Pharmacodynamic |
| PK | pharmacokinetic |
| RNA | ribonucleic acid |
| SC | subcutaneously |
| SD | standard deviation |
| $T_{\text{max}}$ | time of maximum concentration (C <sub>max</sub> ) |
| $t_{1/2}$ | terminal half-life |
| V/F | apparent volume of distribution |

## **Change Log**

| Version | Section | Changes |
|---|---|---|
| 02 | Appendix | Deleted example randomization schedule |
| 03 | 5 | Added that 'Subjects who did not complete their treatment (referred to as early termination subjects) will not be included in PK and PD parameter summary calculations.' |
| 03 | 7.3.1,<br>7.3.2 | The descriptive summary for PD parameters is changed from geometric mean to mean. Changes in PD parameter from baseline for placebo and low doses may have negative values and would not allow for calculation of geometric mean. Text describing the primary, secondary, and exploratory PD parameter was updated for clarity. |
| 03 | General | Typographical changes included throughout |

#### 1. Introduction

This document outlines the proposed statistical methods for data analysis on data collected from Protocol 'SCR-007: Pharmacodynamic Biomarkers to Support Biosimilar Development: Clinical Study 2 (PCSK9 Inhibitors – Alirocumab and Evolocumab)'.

#### 2. Study Objectives

#### 2.1. Primary Objective

The primary objective of this study is to report clinical trial operating characteristics for future clinical pharmacology pharmacokinetics (PK) and pharmacodynamics (PD) similarity studies using the different biomarker-based approaches.

#### 2.2. Secondary Objectives

The secondary objectives of this study are:

- 1. To determine the values and variability of PK and PD parameters at four dose levels (i.e., low, intermediate low, intermediate high, and high doses) for alirocumab and evolocumab.
- 2. Explore PK/PD relationships using appropriate models for alirocumab and evolocumab.

#### 2.3. Exploratory Objective

The exploratory objectives of this study are:

- 1. To evaluate the utility of circulating proteins and small RNAs as potential PD biomarkers.
- 2. To inform analytical approaches and experimental designs needed for identifying exploratory proteomic- and small RNA-based PD biomarkers in plasma

#### 3. Study Overview

#### 3.1. Study Design

This is a randomized, double-blind, placebo-controlled, single-dose, parallel arm, pilot study. Healthy subjects will be randomized to one of four dose groups (low, intermediate low, intermediate high, and high) for each drug (evolocumab or alirocumab) or placebo (See Table 1). The study will be conducted at one center in the United States (Spaulding Clinical Research unit in West Bend, Wisconsin).

U.S. Food and Drug Administration Statistical Analysis Plan: SCR-007

All subjects will be sampled daily for the first week. Subjects in groups A, B, E, and F will follow the schedule of events through day 42. Subjects in groups C and G will follow the schedule of events through day 56. Subjects in groups D, H, and I will follow the schedule of events through day 84. Each treatment group should include equal representation of male and female subjects.

**Table 1: Study Treatment Groups** 

| Subjects (n) | Treatment Group | Drug |
|--------------|-----------------|--------------------------------------------|
| 8 | A | Evolocumab low (21 mg) subcutaneously (SC) |
| 8 | В | Evolocumab intermediate low (35 mg) SC |
| 8 | С | Evolocumab intermediate high (70 mg) SC |
| 8 | D | Evolocumab high (140 mg) SC |
| 8 | Е | Alirocumab low (15 mg) SC |
| 8 | F | Alirocumab intermediate low (25 mg) SC |
| 8 | G | Alirocumab intermediate high (50 mg) SC |
| 8 | Н | Alirocumab high (100 mg) SC |
| 8 | I | Placebo SC |

#### 3.2. Sample size

Approximately 86 healthy subjects will be enrolled (72 subjects for treatment and up to 14 potential replacement subjects). Subjects will be randomized to one of 8 different active treatment arms (i.e. 8 per treatment arm) or placebo. This study did not have any formal sample size or power calculations. Doses expected to characterize the dynamic range of the primary PD parameter (LDL-C) were selected. A total of 8 subjects are planned per dose as a typical sample size for estimating values and variability of PK and PD measures in single ascending dose trials.

#### 4. Study Endpoints

#### 4.1. Primary Endpoints

- Peripheral blood low density lipoprotein-C (LDL-C) area under the effect curve from time zero to last on-study timepoint (AUEC<sub>0-t</sub>, referred to as AUEC for brevity).
- Maximum decrease from baseline in LDL-C (ΔLDL-C<sub>min</sub>)

#### 4.2. Secondary Endpoints

- Area under the curve (AUC) of evolocumab and alirocumab from time zero to infinity (AUC<sub>0-inf</sub>)
- Maximum concentration (C<sub>max</sub>) of evolocumab and alirocumab
- Peripheral blood apolipoprotein B-100 (ApoB) AUEC<sub>0-t</sub>.
- Maximum decrease from baseline in ApoB (ΔApoB<sub>min</sub>)
- Model parameter estimates for evolocumab and alirocumab exposure-response models (exposure parameter versus AUEC<sub>0-t</sub> or ΔLDL-C<sub>min</sub>)

#### 4.3. Exploratory Endpoints

- Peripheral blood proprotein convertase subtilsin/kexin type 9 (PCSK9) AUEC<sub>0-t</sub>.
- Maximum decrease from baseline in PCSK9 (ΔPCSK9<sub>min</sub>)
- Additional pharmacokinetic parameters for evolocumab and alirocumab, including time of maximum concentration (T<sub>max</sub>), elimination rate constant (K<sub>el</sub>), area under the curve from time 0 to end of study (AUC<sub>0-t</sub>), half-life (t<sub>1/2</sub>), apparent clearance (CL/F), and apparent volume of distribution (V/F).
- Time course profiles, maximum increase/decrease from baseline, and AUEC for plasma proteomics and small RNA transcriptomics (set of markers be determined)

#### 5. Analysis Populations

- For all analyses, subjects will be analyzed according to the dose and treatment received,
   not the dose and treatment to which subjects were randomized.
- Subjects who discontinued from the study before their assigned end of study day
   (referred to as early termination subjects) will be excluded from pharmacokinetic and
   pharmacodynamic parameter summary calculations.
- The PD population will include all subjects who receive study drug and have at least 1 estimable PD parameter after dosing. For baseline-adjusted analyses, subjects must also have at least one valid baseline sample between screening to dose administration on day 1. Subjects without a valid baseline sample will be excluded from PD assessments where the derived metric is baseline adjusted.

- The PK population will include all subjects who receive study drug and have at least 1 estimable PK parameter after dosing. Subjects with all samples below the lower limit of quantification will not be included in PK population summaries.
- The PK/PD population (exposure-response population) will include all subjects from the PK and PD populations, including subjects treated with placebo or subjects where all PK samples were below the lower limit of quantification. The PK/PD population will be used for the model-based exposure-response analysis.
- The safety population will include all subjects who receive at least 1 dose of any of the study drugs.

#### 6. Data Screening and Acceptance

#### 6.1. Handling of Missing and Incomplete Data

The following imputation of missing values will be done:

- Pharmacokinetic measurements below the quantification limits will be considered equal to zero for all analyses.
- Non-pharmacokinetic measurements (e.g., LDL-C, ApoB, PCSK9) below the quantification limits will be considered equal to the lower limit of quantification for all analyses unless explicitly noted otherwise.
- Missing pharmacokinetic or pharmacodynamic data (e.g., skipped out patient visit) will not be imputed.
- For baseline adjusted measures, samples from Day 1, time 0 will be used for calculating this derived metric. In cases where the Day 1, time 0 sample is missing or invalid, the sample collected at check-in (Day -1) will be used, followed by the screening sample. If none of these samples are available or valid, then no baseline value will be calculated for the subject.

#### 7. General Statistical Considerations

All data will be presented in data listings. Data from subjects excluded from the analysis population will be presented in the data listings, but not included in the calculation of summary statistics.

#### 7.1. Subject Disposition

The number of subjects who enroll in the study and the number and percentage of subjects who complete each assessment will be presented. The frequency and percentage of subjects who withdraw or discontinue from the study and the reason for withdrawal or discontinuation will be summarized. In addition, significant known protocol deviations will be noted for individual subjects.

#### 7.2. Demographics and Baseline Characteristics

Descriptive statistics will be used to summarize demographic and baseline subject characteristics for age, sex, weight, body mass index, race, and ethnicity. For continuous variables, the mean, median, standard deviation (SD), minimum, and maximum values will be reported. For categorical (nominal) variables, the number and percentage of subjects (or observations) will be reported.

#### 7.3. Pharmacodynamic Analysis

#### 7.3.1 LDL-C

Individual LDL-C versus time plots will be presented for each participant. For LDL-C, AUEC and maximum decrease from baseline will be calculated for each participant using all on treatment timepoints. Calculations will be performed using non-compartmental analysis packages available in statistical software. The primary analysis with LDL-C will use baseline adjusted AUEC and maximum decrease from baseline; other derived AUEC measures may be calculated (AUEC calculation without baseline adjustment and with normalization to baseline [pAUEC]) to evaluate how derived PD metrics impact trial design. PD parameters of evolocumab, alirocumab, and placebo groups will be listed and summarized using descriptive statistics (n, mean, SD, coefficient of variation, minimum, median, interquartile range, and maximum) for each treatment arm.

#### 7.3.2 ApoB and PCSK9

Individual ApoB and PCSK9 versus time plots will be presented for each participant. For ApoB and PCSK9, baseline-adjusted AUEC and maximum decrease from baseline will be calculated for each participant using all on treatment timepoints. Calculations will be performed using non-compartmental analysis packages available in statistical software. The secondary analysis with ApoB will use baseline adjusted AUEC and maximum decrease from baseline. The exploratory analysis with PCSK9 will use baseline adjusted AUEC and maximum decrease from baseline. Other derived AUEC measures for ApoB and PCSK9 may be calculated (AUEC calculation without baseline adjustment and with normalization to

baseline [pAUEC]) to evaluate how derived PD metrics impact trial design. PD parameters of evolocumab, alirocumab, and placebo groups will be listed and summarized using descriptive statistics (n, mean, SD, coefficient of variation, minimum, median, interquartile range, and maximum) for each treatment arm.

#### 7.4. Pharmacokinetic Analysis – Alirocumab and Evolocumab

Individual serum concentration versus time plots for evolocumab and alirocumab groups will be presented for each participant. AUC<sub>0-inf</sub> and C<sub>max</sub> will be calculated for each participant using all on treatment timepoints as part of the secondary analysis. In addition, the following PK parameters will be calculated for each individual as exploratory analyses: AUC<sub>0-t</sub>, T<sub>max</sub>, apparent clearance (CL/F), apparent volume of distribution (V/F), elimination rate (Kel), and terminal half-life (t<sub>1/2</sub>) PK parameters will be calculated for each participant using all on treatment timepoints. All parameters will be summarized using descriptive statistics (n, geometric mean, coefficient of variation, minimum, median, interquartile range, and maximum) for each alirocumab and evolocumab treatment arm.

Calculations will be performed using non-compartmental analysis packages available in statistical software. Serum concentrations below the limits of quantification will be set to zero for the purpose of this analysis. Subjects with all samples below the limit of quantification will be excluded from PK summaries.  $AUC_{0-inf}$ ,  $t_{1/2}$ , and Kel for subjects will only be included for subjects with 3 or more concentration values on the terminal portion of the pharmacokinetic curve and with an adjusted coefficient of determinations ( $R^2$ ) greater than 0.80.

#### 7.5. PK/PD Analyses

The dose- and exposure-response relationship between baseline-adjusted AUEC for LDL-C and  $\Delta$ LDL-C<sub>min</sub> and alirocumab and evolocumab will be explored graphically (separate assessments for both response measures). Based on these observations, model-based analyses using statistical software will be conducted separately for each drug with respect to each of the above-mentioned PD measures.

The model-based analysis will explore both dose and exposure (i.e., AUC<sub>0-inf</sub>, referred to as AUC below) as the dependent variable. All dose levels for a drug, as well as placebo data, will be

U.S. Food and Drug Administration Statistical Analysis Plan: SCR-007

combined for the analysis. Model selection will be based on the initial graphical assessment and will be selected from one of the following structures – linear,  $E_{max}$ , and sigmoidal. Multiple models may be evaluated based on the initial graphical analysis, in which case model selection will be based on a combination of goodness of fit plots, parameter uncertainty (i.e., parameter confidence intervals including zero), and Akaike's information criterion (AIC). General representations for each of the model structures and parameterizations is shown below:

#### Dose-relationship

Linear: Response  $\sim E_0 + \text{Slope * Dose}$ 

 $E_{\text{max}}$ : Response ~  $E_0 + E_{\text{max,dose}} * Dose / (Dose + ED_{50})$ 

Sigmoidal: Response  $\sim E_0 + E_{\text{max,dose}} * \text{Dose}^{\gamma} / (\text{Dose}^{\gamma} + \text{ED}_{50}^{\gamma})$ 

#### Exposure-relationship

Linear: Response  $\sim E_0 + \text{Slope * AUC}$ 

 $E_{max}$ : Response ~  $E_0 + E_{max,exp} * AUC / (AUC + EC_{50})$ 

Sigmoidal: Response  $\sim E_0 + E_{max,exp} * AUC^{\gamma} / (AUC^{\gamma} + EC_{50}^{\gamma})$ 

Model evaluation will include residual variability error term but will not include any random effects or covariate evaluation on fixed effect.

#### 7.6. Exploratory Omics Analysis

Various proteomics, transcriptomics, and genomic analyses may be performed on collected data for biomarker exploration. Additional details regarding the statistical methods for these analyses will be described in a separate plan.

#### 7.7. Safety Analyses

#### 7.7.1 Adverse Events

All AEs will be coded using the latest version of the Medical Dictionary for Regulatory Activities. The incidence of TEAEs, organized by system organ class and frequency, will be summarized by seriousness, severity, relationship to treatment, and by treatment at onset of the TEAE. A detailed listing of serious AEs and TEAEs leading to withdrawal will also be provided.

#### 7.7.2 Clinical Laboratory Tests

Clinical laboratory results (hematology, serum chemistry, and urinalysis) will be summarized using descriptive statistics (number of subjects, mean, SD, minimum, median, and maximum). Clinical laboratory results will be classified as normal or abnormal, according to the reference ranges of the individual parameter. No statistical testing will be performed on clinical laboratory data.

#### 7.7.3 Vital Sign Measurements

Vital sign measurements and changes from Baseline will be summarized using descriptive statistics (number of subjects, mean, SD, minimum, median, and maximum) by treatment and time point.

#### 7.7.4 Safety 12-lead Electrocardiograms

The incidence of pathological ECG interpretive statements at Baseline and during treatment will be assessed among the treatments.

#### 7.7.5 Physical Examinations

Physical examination findings will be presented in a data listing, and abnormal physical examination findings will be recorded as AEs.

#### 7.7.6 Other Safety Data

All concomitant medication usage and medications that changed in daily dose, frequency, or both since the subject provided informed consent will be summarized for each subject.

#### 8. Data Quality Assurance

Completed eCRFs are required for each subject randomly assigned to study drug. Electronic data entry will be accomplished through the ClinSpark® remote electronic data capture system, which allows for on-site data entry and data management. This system provides immediate, direct data transfer to the database, as well as immediate detection of discrepancies, enabling site coordinators to resolve and manage discrepancies in a timely manner. Each person involved with the study will have an individual identification code and password that allows for record traceability. Thus, the system, and subsequently any investigative reviews, can identify coordinators, investigators, and individuals who have entered or modified records.

Furthermore, the investigator retains full responsibility for the accuracy and authenticity of all data entered into the electronic data capture system. The completed dataset and their associated files are the sole property of the sponsor and should not be made available in any form to third parties, except for appropriate governmental health or regulatory authorities, without written permission of the sponsor.

## Attachment A. Pharmacokinetic, Pharmacodynamic, and Biomarker Sample Collection Schedule

#### **Pharmacokinetic Sample Collection**

Pharmacokinetic blood samples (5 mL) for determination of evolocumab or alirocumab concentration will be collected at the following time points:

- Day 1: 0 (pre-dose), 0.5, 1, 2, 3, 4, 6, 8, 12, 24 h
- Day 2, 3, 4, 5, 6, 7, 10, 14, 21, 28, 35, 42, 56, 70, 84

Blood samples will be collected by direct venipuncture or by inserting an IV catheter into the subject's forearm region. Each blood sample will be labeled with subject number, study number, study day, time point, event, and a barcode that matches that belonging to the subject.

#### **Pharmacodynamic Sample Collection**

Blood samples (5 mL) for primary pharmacodynamic biomarker (peripheral blood LDL-C) and secondary pharmacodynamic biomarker (peripheral blood ApoB) assessment will be collected at the following time points:

- Screening (Day -21 to -2)
- Day -1 (check-in)
- Day 1: 0 (Pre-dose) and 24 h (Day 2)
- Day 3, 4, 5, 7, 10, 14, 21, 28, 35, 42, 56, 70, 84

Blood samples will be collected by direct venipuncture or by inserting an IV catheter into the subject's forearm region. Each blood sample will be labeled with subject number, study number, study day, time point, event, and a barcode that matches that belonging to the subject.

#### **Exploratory PD Biomarkers**

Exploratory PD biomarkers will be evaluated using plasma proteomics and small RNA transcriptomics. Whole blood samples (5 mL) will be collected and processed for plasma at the following time points:

- Day -1 (check-in)
- Day 1: 0 (pre-dose), 0.5, 1, 2, 3, 4, 6, 8, and 12 h; 24 h (Day 2)
- Day 3, 4, 5, 6, 7, 7, 10, 14, 21, 28, 35, 42, 56, 70, 84

Blood samples will be collected by direct venipuncture or by inserting an IV catheter into the subject's forearm region. Each blood sample will be labeled with subject number, study number,

study day, time point, event, and a barcode that matches that belonging to the subject. All blood samples will be processed for preparation of plasma.

#### **Attachment B. Randomization Schedule**

Subjects will enter the study clinic for check-in procedures the day before study drug administration of the first period (Day -1). All study drugs will be administered subcutaneously. On Day 1, subjects will receive their assigned treatment according to the randomization schedule generated by the project biostatistician and provided to designated unblinded recipients (i.e., pharmacist) at the clinical site.

| Treatment Group | Drug |
|-----------------|--------------------------------------|
| A | Evolocumab low (21 mg) |
| В | Evolocumab intermediate low (35 mg) |
| С | Evolocumab intermediate high (70 mg) |
| D | Evolocumab high (140 mg) |
| Е | Alirocumab low (15 mg) |
| F | Alirocumab intermediate low (25 mg) |
| G | Alirocumab intermediate high (50 mg) |
| Н | Alirocumab high (100 mg) |
| I | Placebo |